CLINICAL TRIAL: NCT02105519
Title: The Immunogenicity and Safety of the Seasonal Influenza Vaccine, Formulation 2013-2014, in Chronic Kidney Disease Patients Not on Dialysis
Brief Title: The Effect and Safety of the Seasonal Trivalent Influenza Vaccine in Chronic Kidney Disease Patients Not on Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Tzu Chang, Attending physician, National Cheng-Kung University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-101-139
Record Dates: First submitted 2013-12-09; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Immunogenicity and Adverse Drug Effect of Vaccines Influenza; Chronic Kidney Disease
Keywords: trivalent influenza vaccine, chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- The group receiving no influenza vaccine (No Intervention): Participants in this group will not receive any influenza vaccine (negative control group).
- One dose of AdimFlu-S group (Experimental): Participants in this group will receive one dose of the seasonal trivalent influenza vaccine (one dose of AdimFlu-S group), formulation 2013-2014, at the initiation of the study. Each administered dose contain 15 ug virus antigen for each virus strain.
  Interventions: Biological: Seasonal influenza vaccine (AdimFlu-S)
- Two dose of AdimFlu-S group (Experimental): Participants in this group (Two dose of AdimFlu-S group)will receive the seasonal trivalent influenza vaccine, formulation 2013-2014, at the week 0 and 4 weeks after the initiation of the study. Each administered dose contain 15 ug virus antigen for each virus strain.
  Interventions: Biological: Seasonal influenza vaccine (AdimFlu-S)

INTERVENTIONS:
Biological: Seasonal influenza vaccine (AdimFlu-S) — Participants receiving 0, 1 and 2 dose of AdimFlu-S during the study period.(a) No vaccination: no any influenza vaccination during the study period.(b) One dose of AdimFlu-S group: patient will receive one dose of Seasonal influenza vaccine (AdimFlu-S) at the initiation of the study.(c)Two doses of AdimFlu-S group: patients will receive one dose of Seasonal influenza vaccine (AdimFlu-S) at week 0 and 4 weeks after the initiation of the study.
  Other Names: AdimFlu-S, manufactured by Adimmune company.
  Arms: One dose of AdimFlu-S group; Two dose of AdimFlu-S group

SUMMARY:
In recent years, several studies revealed that the current influenza vaccine strategy might be of minimal vaccine effectiveness and had a smaller effect on reducing morbidity and mortality in the end-stage renal disease population than previously thought. Thus, this also raised the question about the effectiveness of administration of influenza vaccination in chronic kidney disease patients not on dialysis. In this study, the investigators aim to evaluate the effectiveness of seasonal trivalent influenza vaccine, formulation 2013-2014, in patients with different stage of chronic kidney disease (CKD) not on dialysis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the antibody response to each of the three influenza vaccine strains included in the licensed seasonal flu vaccine, as measured by the method of hemagglutination inhibition (HI) and ELISA-based microneutralization (microNT-ELISA) assays. All participants will be divided into 3 groups: participants refused to receive vaccination, those receive either one (week 0) or one more booster vaccination (week 0 and week 4). The investigators will collect serum of participants at the 5th weeks, 9th weeks, and 21th week post vaccination and evaluate the difference of immune response in these 3 groups.

ELIGIBILITY:
Inclusion Criteria:

1. .Males and non-pregnant females and aged ≥ 18 years with chronic kidney disease not on dialysis;
2. .Willing and able to adhere to visit schedules and all study requirements;
3. .Subjects read and signed the study-specific informed consent.
4. .Subjects who has either received the first dose of 2013-2014 seasonal influenza vaccination before or not.

Exclusion Criteria:

1. .Subject or his/her family is employed by the participated hospital;
2. .History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication;
3. .Personal or family history of Guillain-Barré Syndrome;
4. .An acute febrile illness within 1 week prior to vaccination;
5. .Current upper respiratory illness, including the common cold or nasal congestion within 72 hours;
6. .Subjects with influenza-like illness as defined by the presence of fever (temperature ≥ 38°C) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
7. .Female subjects who are pregnant during the study.
8. .Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
9. .Immunodeficiency, or under immunosuppressive treatment.
10. .Receipt of any vaccine within 1 week prior to study vaccination or expected receipt between Visit 1 (study vaccination) and Visit 2 (final collection of blood samples);
11. .Receipt of any blood products, including immunoglobulin in the prior 3 months;
12. .Any severe illness needed to be hospitalization within three months.
13. .Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The dynamic change of seroprotection rate related to administration of influenza virus vaccine strains (2013-2014 season) of the AdimFlu-S manufactured by Adimmune Corporation. | The seroprotection rate will be assessed at 4, 8, 20 weeks after the initiation of the study.
  The primary endpoint will be the seroprotection rate which is defined as the proportion of subjects with HI titer ≥ 1:40. MicroNT-ELISA assay might also be used to evaluate the seroprotection post vaccination, which will be defined as micro-NT titer ≥1: 40 or ≥ 1:160 .

SECONDARY OUTCOMES:
The safety of the influenza vaccination in patients with chronic kidney disease. | the safety issue related to the vaccination will be assessed in each visit during the whole study period (20 weeks).
  Patients who received influenza vaccination would be asked to record any local or systemic side effect during the first week after vaccination. Besides, the investigators would also monitor any possible adverse effect during the whole study period.
The dynamic change of seroconversion rate related to administration of influenza virus vaccine strains (2013-2014 season) of the AdimFlu-S manufactured by Adimmune Corporation. | The seroconversion rate will be assessed at 4, 8, 20 weeks after the initiation of the study.
  The seroconversion is defined as the HI titer of the post-vaccination serum is at least 1:40 for those who had a negative pre-vaccination HI serum titer or a four-fold or greater increase in HI titers in subjects who had a positive pre-vaccination HAI serum titer. The seropositive is defined as the HI titer ≥ 1:10, and the seronegative is defined as HI titer < 1:10.
The dynamic change of seroresponse rate related to administration of influenza virus vaccine strains (2013-2014 season) of the AdimFlu-S manufactured by Adimmune Corporation. | The seroresponse rate will be assessed at 4, 8, 20 weeks after the initiation of the study.
  The seroresponse is defined as HI or micro-NT titer of the post-vaccination serum is at least 4-fold increase of the HI or micro-NT titer after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheng Wang, MD, Principal Investigator — National Cheng Kung University and Hospital; Chin-Chung Tseng, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital; Junne-Ming Sung, MD, Principal Investigator — National Cheng Kung University and Hospital; An-Bang Wu, MD, Principal Investigator — National Cheng-Kung University Hospital; Wei-Hung Lin, ＭＤ, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University, Tainan, Taiwan, Taiwan